CLINICAL TRIAL: NCT06932484
Title: A NEW APPROACH IN THE MANAGEMENT OF INTRAOPERATIVE ARTERIAL HYPOTENSION BASED ON DELTA VARIATION OF HEMODYNAMIC PARAMETERS: A RANDOMISED CLINICAL TRIAL
Brief Title: Delta Variation to Guide Hemodynamic Optimization
Acronym: DELTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RUSSO ANDREA, MD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7428
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Hemodynamic MAP Stability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- delta (Experimental): in this group the trigger for any intervention will be the delta variation of the hemodynamic parameters showed in the monitoring platform
  Interventions: Procedure: parameters
- standard (No Intervention): in this group hemodynamics will be managed by using the hypotension prediction index

INTERVENTIONS:
Procedure: parameters — during surgery hemodynamic will be optimized based on percentage variation of different variables
  Arms: delta

SUMMARY:
intraoperative hemodynamic optimization will be based on the percentage of variation of the parameters

ELIGIBILITY:
Inclusion Criteria: All patients > 18 years old scheduled for major abdominal

Exclusion Criteria:

Body Mass Index > 35 kg/m2 Pregnancy Refusal to sign written informed consent Urgent and/or emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
time weighted average of mean arterial pressure | the end of surgery
  we will avoid hypotensive episodes by using a predictive approach and then calculate the TWA-MAP < 65 mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided